CLINICAL TRIAL: NCT07354867
Title: Effect of Simplified Robot (FASTER) Assisted Versus Conventional Endoscopic Submucosal Dissection (ESD) for Colorectal Lesions: A Prospective, Randomized, Controlled Trial
Brief Title: Effect of Simplified Robot (FASTER) Assisted Versus Conventional Endoscopic Submucosal Dissection (ESD) for Colorectal Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiyun Liu (Other)
Responsible Party: Sponsor-Investigator, Kaiyun Liu, Principal Investigator, Clinical Professor, Shenzhen Hospital of Southern Medical University
Organization: Shenzhen Hospital of Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYSZYYEC2025K111R002
Record Dates: First submitted 2026-01-04; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Lesions; Endoscopic Submucosal Dissection (ESD); FASTER Robot
Keywords: Endoscopic Submucosal Dissection (ESD); Colorectal lesions; FASTER robot; Procedure time; Randomized controlled trial (RCT)

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups: a FASTER robot-assisted ESD group or a conventional ESD group. Both groups will undergo the assigned endoscopic submucosal dissection procedure for colorectal lesions performed by experienced endoscopists. In the robot-assisted group, the FASTER robotic arm will provide multidirectional traction using its end-effector grasper to optimize the submucosal field during dissection, whereas the control group will complete submucosal dissection using standard ESD techniques. Outcomes will be compared between groups to evaluate differences in procedure time, mucosal dissection time and speed, resection quality, complication rates, procedural stability, and robotic maneuverability.
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study in which the outcomes assessor is blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FASTER robot-assisted ESD group (Experimental): FASTER robot-assisted ESD group - Patients undergo ESD with the FASTER robotic arm attached to the endoscope tip, with robotic grasping to assist submucosal dissection.
  Interventions: Other: FASTER robot-assisted ESD group
- Conventional colorectal ESD (Active Comparator): Conventional colorectal ESD - Patients undergo standard ESD using a transparent distal cap without robotic assistance.
  Interventions: Other: Conventional ESD group

INTERVENTIONS:
Other: FASTER robot-assisted ESD group — In the experimental group, the FASTER robotic arm will be attached to the tip of the endoscope at the beginning of the procedure. ESD will then be performed according to the standard steps of conventional ESD: (1) lesion marking; (2) submucosal injection with normal saline mixed with indigo carmine; and (3) circumferential incision. After completion of the submucosal injection and circumferential incision, the robotic arm will be deployed, and the end-effector grasper will grasp and lift the mucosal edge to provide a clear view of the dissection plane, after which submucosal dissection will be performed. Finally, the resected specimen will be retrieved using the FASTER system through the endoscope or via suction. Throughout the procedure, patients' vital signs and any procedure-related serious adverse events will be recorded for statistical analysis
  Arms: FASTER robot-assisted ESD group
Other: Conventional ESD group — In the control group, a transparent distal attachment cap will be mounted onto the tip of the endoscope at the beginning of the procedure. ESD will then be performed following the standard steps of conventional ESD, including: (1) lesion marking; (2) submucosal injection using normal saline mixed with indigo carmine; (3) circumferential incision; (4) submucosal dissection; and (5) retrieval of the resected specimen via suction. Throughout the procedure, patients' vital signs and any procedure-related serious adverse events will be recorded for statistical analysis.
  Arms: Conventional colorectal ESD

SUMMARY:
This study aims to compare the outcomes of Simplified Robot (FASTER) assisted Endoscopic Submucosal Dissection (ESD) with conventional ESD in the treatment of colorectal lesions. Using a prospective, single-center, randomized controlled design, the investigators will systematically evaluate differences between the two approaches in terms of total procedure time, mucosal dissection time and speed, resection quality (R0 resection rate and en bloc resection rate), incidence of complications (bleeding, perforation, muscularis injury), and the flexibility and clinical feasibility of robotic operation. The clinical significance of this study lies in assessing the value of robotic assistance in colorectal ESD, optimizing intraoperative workflow, reducing complication risks, improving patient outcomes and procedural efficiency, and providing evidence to support individualized therapeutic strategies in clinical practice.This study aims to compare the outcomes of Simplified Robot (FASTER) assisted Endoscopic Submucosal Dissection (ESD) with conventional ESD in the treatment of colorectal lesions. Using a prospective, single-center, randomized controlled design, the investigators will systematically evaluate differences between the two approaches in terms of total procedure time, mucosal dissection time and speed, resection quality (R0 resection rate and en bloc resection rate), incidence of complications (bleeding, perforation, muscularis injury), and the flexibility and clinical feasibility of robotic operation. The clinical significance of this study lies in assessing the value of robotic assistance in colorectal ESD, optimizing intraoperative workflow, reducing complication risks, improving patient outcomes and procedural efficiency, and providing evidence to support individualized therapeutic strategies in clinical practice.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized controlled trial enrolling patients scheduled to undergo endoscopic submucosal dissection (ESD) for colorectal lesions. Eligible subjects will be screened according to predefined inclusion and exclusion criteria and, after providing written informed consent, randomized 1:1 to the experimental group (FASTER robot-assisted ESD) or the control group (conventional ESD). All participants will undergo standardized ESD performed by experienced endoscopists.

In the experimental group, after a circumferential incision is completed, the FASTER robotic arm will be used; its end-effector grasper will apply multidirectional traction to the lesion margins to optimize the submucosal field before completing the dissection. The control group will undergo mucosal-submucosal dissection using conventional ESD techniques.

Postoperatively, all participants will receive routine acid-suppression therapy and begin a warm, cool liquid diet 6 hours after the procedure. If no intolerance occurs within 24 hours, the diet will be advanced stepwise to semi-liquid and then soft foods until discharge.

During treatment, the following parameters will be recorded and evaluated: total procedure time, mucosal dissection time and dissection speed, resection quality (R0 resection rate and en-bloc resection rate), complication rates (bleeding, perforation, muscularis propria injury), procedural stability, and robotic maneuverability. All participants will be followed during the postoperative hospitalization period, with collection of clinical status, laboratory results, and device-related information.

The study team will conduct statistical analyses to compare the two approaches in terms of efficacy and safety, evaluate their clinical applicability, and provide scientific evidence to support optimization of colorectal ESD workflows and the broader adoption of robot-assisted technology.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Patients with colorectal lesions scheduled to undergo endoscopic submucosal dissection (ESD)
3. Lesion characteristics meeting any of the following criteria: (1) Lesions unsuitable for en bloc resection using snare-based EMR, including non-granular type laterally spreading tumors (LST-NG), especially pseudo-depressed subtype (PD); lesions with type VI pit pattern (VI-type glandular opening configuration); carcinomas with superficial submucosal invasion (T1-SM); large depressed-type tumors; large protruding lesions suspected of malignancy, including nodular mixed-type granular LSTs (LST-G); other lesions unsuitable for en bloc resection using snare-based EMR; (2) Lesions with special background conditions, including mucosal tumors with submucosal fibrosis (caused by prior biopsy or mucosal prolapse due to peristalsis); sporadic tumors arising in the context of chronic inflammation (e.g., ulcerative colitis); local residual or recurrent early carcinoma following prior endoscopic resection;
4. Willingness to participate in the study and provision of written informed consent.

Exclusion Criteria:

1. Suspected deep submucosal invasive carcinoma based on endoscopic features；
2. Lesions presenting with non-lifting signs, suggesting deep submucosal invasive carcinoma or tumors with severe submucosal fibrosis;
3. Lesions extending to the appendiceal orifice, colonic diverticulum, or ileocecal valve; (4) Pregnant women or women who may be pregnant; lactating women;
4. Pregnant women or women who may be pregnant; lactating women;
5. Patients with coagulation disorders;
6. Patients considered ineligible for specific reasons;
7. Patients with contraindications to anesthesia and/or colonoscopy. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Total procedure time | Recorded intraoperatively
  Measured from initiation of submucosal injection to completion of submucosal dissection.

SECONDARY OUTCOMES:
En bloc resection rate | Periprocedural (intraoperative assessment)
  Defined as whether the lesion was resected in a single piece, assessed immediately after resection by the endoscopist.
Submucosal dissection time | Recorded intraoperatively
  Measured from completion of circumferential incision to complete removal of the lesion
Robotic operational flexibility | Recorded intraoperatively
  Number of attempts required for successful grasp and number of accidental drops. Successful grasp defined as effective traction providing clear submucosal visualization.
Dissection speed | Periprocedural (from intraoperative measurement to postoperative calculation within 24 hours)
  Calculated as lesion area divided by dissection time. Lesion area is determined intraoperatively or from the resected specimen using the longest diameter (a) and the perpendicular diameter (b), applying the ellipse formula: area = a × b × π/4.
Incidence of device malfunction | Recorded intraoperatively
  Device malfunctions (arm jamming, vision interruption, waterway obstruction/leakage) will be recorded intraoperatively and expressed as events per total cases.
Rates of intraoperative and postoperative complications | Periprocedural (from intraoperative period through hospital discharge, up to 7 days)
  Intraoperative and postoperative complications such as bleeding, perforation, and muscularis propria injury will be documented. Based on established clinical diagnostic criteria and the corresponding medical records, these events will be assessed by the study investigators and recorded in the CRF.
Complete resection rate | Within 7 days post-procedure (upon pathology report issuance)
  Defined as en bloc resection with histologically tumor-free lateral and vertical margins (R0 resection).

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT07354867/Prot_SAP_000.pdf